CLINICAL TRIAL: NCT06883591
Title: Physical Activity in Patients After Resurfacing and Total Hip Arthroplasty: an Observational Follow-up Study 15 Years After Surgery.
Brief Title: Triaxial Accelerometry Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-2605; 2025-17970 (Other: METC Oost-Nederland)
Record Dates: First submitted 2025-03-05; First posted 2025-03-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Total Hip Arthroplasty (THA); Accelerometers; Resurfacing Hip Arthroplasty
Keywords: Total Hip Arthroplasty; Observation; Accelerometry; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Resurfacing Hip Arthroplasty: Patients 15 years after hip resurfacing surgery
- Total Hip Arthroplasty: Patients 15 years after Total Hip Arthroplasty

SUMMARY:
This study looks at how physical activity levels are in the long term after hip surgery. Arthritis can make everyday movement difficult, and hip replacement surgeries-such as total hip arthroplasty (THA) and hip resurfacing-help reduce pain and improve function. However, it is not clear how these surgeries affect long-term physical activity.

To learn more, researchers are following up with patients who had one of these surgeries 15 years ago. Participants will wear two small activity-tracking devices (accelerometers): one on their wrist for 10 days and one on their thigh for 48 hours. These devices will measure how much and how intensely they move. Participants will also complete short physical activity questionnaires.

By comparing activity levels between the two types of hip surgery, the study aims to understand their long-term effects on mobility and health. The results could help doctors improve treatment and recovery plans for future patients. All data will be kept private, and participation is voluntary.

DETAILED DESCRIPTION:
Arthritis significantly impacts patients' quality of life, leading to pain, fatigue, and reduced mobility. Treatment strategies include medication, lifestyle changes, and surgical interventions such as total hip arthroplasty (THA) and hip resurfacing. While these procedures improve function and alleviate pain, their long-term effects on physical activity levels remain unclear. Given the importance of physical activity in maintaining health and reducing mortality risks, understanding post-surgical activity levels is crucial.

Wearable technology has revolutionized the measurement of physical activity, providing objective, large-scale data collection. This study utilizes accelerometers to evaluate physical activity in patients who underwent hip resurfacing or THA 15 years ago. By comparing these groups, researchers aim to understand the long-term impact of different surgical interventions on mobility and activity levels.

The primary objective of the study is to compare the volume and intensity of physical activity in patients who underwent hip resurfacing versus those who had a total hip replacement. We will also explore associations between physical activity levels and functional outcome scores.

This is a cross-sectional observational study involving a follow-up of patients who participated in a randomized controlled trial 15 years ago. Participants will be asked to complete questionnaires and wear two different accelerometers to monitor their physical activity. They will wear a GENEActiv triaxial accelerometer on the non-dominant wrist for 10 days and nights. They will also wear an Axivity AX3 Logging triaxial accelerometer on the surgical thigh for 48 hours. Both will measure physical activity energy expenditure (PAEE), intensity distribution of PAEE, and step count.

All participants will receive an information letter and provide informed consent before participation. Data privacy will be maintained through coded identifiers, and no personally identifiable information will be stored with the accelerometry data.

This study will provide valuable insights into the long-term mobility outcomes of patients who have undergone hip resurfacing or total hip arthroplasty. The findings will help clinicians understand the implications of surgical choices on patients' activity levels and overall health, potentially influencing future treatment recommendations and rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

• Patient must have participated in a previous randomised controlled trial that was conducted in Rijnstate hospital between 2007-2008.

Exclusion Criteria:

• None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have previously participated in a randomised controlled trial during which they received either hip resurfacing or total hip arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective physical activity | Physical activity measured continuously for a duration of 10 days
  Physical activity energy expenditure (PAEE) and physical activity intensity distribution as measured by two accelerometers

SECONDARY OUTCOMES:
Self-reported physical activity | Seven days prior to the first day of accelerometer use
  Self-reported physical activity using a Dutch version of the International Physical Activity Questionnaire - Short Form (IPAQ-SF).
Self-reported physical activity | Seven days prior to the first day of accelerometer use
  Self-reported physical activity using a Dutch version of the Short Questionnaire to Assess health-enhancing physical activity (SQUASH).

OTHER OUTCOMES:
Step count | Daily steps taken over a period of 10 days
  The participants' daily number of steps taken as measured by two accelerometers

CONTACTS AND LOCATIONS:
Overall Officials: Job LC Susante, MD, PhD, Principal Investigator — Stichting Rijnstate Ziekenhuis
Locations (2):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haverkamp D, Breugem SJ, Sierevelt IN, Blankevoort L, van Dijk CN. Translation and validation of the Dutch version of the Oxford 12-item knee questionnaire for knee arthroplasty. Acta Orthop. 2005 Jun;76(3):347-52. PMID 16156462
- [Background] Wylde V, Learmonth ID, Cavendish VJ. The Oxford hip score: the patient's perspective. Health Qual Life Outcomes. 2005 Oct 31;3:66. doi: 10.1186/1477-7525-3-66. PMID 16259627
- [Background] Dawson J, Fitzpatrick R, Murray D, Carr A. Comparison of measures to assess outcomes in total hip replacement surgery. Qual Health Care. 1996 Jun;5(2):81-8. doi: 10.1136/qshc.5.2.81. PMID 10158596
- [Background] Gosens T, Hoefnagels NH, de Vet RC, Dhert WJ, van Langelaan EJ, Bulstra SK, Geesink RG. The "Oxford Heup Score": the translation and validation of a questionnaire into Dutch to evaluate the results of total hip arthroplasty. Acta Orthop. 2005 Apr;76(2):204-11. doi: 10.1080/00016470510030580. PMID 16097545
- [Background] Stolk E, Ludwig K, Rand K, van Hout B, Ramos-Goni JM. Overview, Update, and Lessons Learned From the International EQ-5D-5L Valuation Work: Version 2 of the EQ-5D-5L Valuation Protocol. Value Health. 2019 Jan;22(1):23-30. doi: 10.1016/j.jval.2018.05.010. Epub 2019 Jan 2. PMID 30661630
- [Background] M Versteegh M, M Vermeulen K, M A A Evers S, de Wit GA, Prenger R, A Stolk E. Dutch Tariff for the Five-Level Version of EQ-5D. Value Health. 2016 Jun;19(4):343-52. doi: 10.1016/j.jval.2016.01.003. Epub 2016 Mar 30. PMID 27325326
- [Background] Devlin N, Roudijk B, Ludwig K, editors. Value Sets for EQ-5D-5L: A Compendium, Comparative Review & User Guide [Internet]. Cham (CH): Springer; 2022. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK589304/ PMID 36810025
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Vandelanotte C, De Bourdeaudhuij I, Philippaerts R, Sjöström M, Sallis J. Reliability and Validity of a Computerized and Dutch Version of the International Physical Activity Questionnaire (IPAQ). Journal of Physical Activity and Health. 2005;2(1):63-75.
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Silsbury Z, Goldsmith R, Rushton A. Systematic review of the measurement properties of self-report physical activity questionnaires in healthy adult populations. BMJ Open. 2015 Sep 15;5(9):e008430. doi: 10.1136/bmjopen-2015-008430. PMID 26373402
- [Background] Kraus WE, Janz KF, Powell KE, Campbell WW, Jakicic JM, Troiano RP, Sprow K, Torres A, Piercy KL; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. Daily Step Counts for Measuring Physical Activity Exposure and Its Relation to Health. Med Sci Sports Exerc. 2019 Jun;51(6):1206-1212. doi: 10.1249/MSS.0000000000001932. PMID 31095077
- [Background] Gerhardt DMJM, Mors TGT, Hannink G, Van Susante JLC. Resurfacing hip arthroplasty better preserves a normal gait pattern at increasing walking speeds compared to total hip arthroplasty. Acta Orthop. 2019 Jun;90(3):231-236. doi: 10.1080/17453674.2019.1594096. Epub 2019 Apr 1. PMID 30931667
- [Background] Maillot C, Auvinet E, Harman C, Cobb J, Riviere C. Hip resurfacing generates a more physiological gait than total hip replacement: A case-control study. Orthop Traumatol Surg Res. 2020 May;106(3):527-534. doi: 10.1016/j.otsr.2019.12.020. Epub 2020 Apr 4. PMID 32265178
- [Background] Garner AJ, Dandridge OW, van Arkel RJ, Cobb JP. Medial bicompartmental arthroplasty patients display more normal gait and improved satisfaction, compared to matched total knee arthroplasty patients. Knee Surg Sports Traumatol Arthrosc. 2023 Mar;31(3):830-838. doi: 10.1007/s00167-021-06773-8. Epub 2021 Oct 23. PMID 34689224
- [Background] Garner AJ, Dandridge OW, van Arkel RJ, Cobb JP. The compartmental approach to revision of partial knee arthroplasty results in nearer-normal gait and improved patient reported outcomes compared to total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2023 Mar;31(3):1143-1152. doi: 10.1007/s00167-021-06691-9. Epub 2021 Aug 20. PMID 34415369
- [Background] NJR. National Joint Registry 8th Annual Report. 2011.
- [Background] Grimes L, Outtrim JG, Griffin SJ, Ercole A. Accelerometery as a measure of modifiable physical activity in high-risk elderly preoperative patients: a prospective observational pilot study. BMJ Open. 2019 Nov 3;9(11):e032346. doi: 10.1136/bmjopen-2019-032346. PMID 31685513
- [Background] Doherty A, Jackson D, Hammerla N, Plotz T, Olivier P, Granat MH, White T, van Hees VT, Trenell MI, Owen CG, Preece SJ, Gillions R, Sheard S, Peakman T, Brage S, Wareham NJ. Large Scale Population Assessment of Physical Activity Using Wrist Worn Accelerometers: The UK Biobank Study. PLoS One. 2017 Feb 1;12(2):e0169649. doi: 10.1371/journal.pone.0169649. eCollection 2017. PMID 28146576
- [Background] Dumuid D, Lewis LK, Olds TS, Maher C, Bondarenko C, Norton L. Relationships between older adults' use of time and cardio-respiratory fitness, obesity and cardio-metabolic risk: A compositional isotemporal substitution analysis. Maturitas. 2018 Apr;110:104-110. doi: 10.1016/j.maturitas.2018.02.003. Epub 2018 Feb 7. PMID 29563028
- [Background] Chastin S, McGregor D, Palarea-Albaladejo J, Diaz KM, Hagstromer M, Hallal PC, van Hees VT, Hooker S, Howard VJ, Lee IM, von Rosen P, Sabia S, Shiroma EJ, Yerramalla MS, Dall P. Joint association between accelerometry-measured daily combination of time spent in physical activity, sedentary behaviour and sleep and all-cause mortality: a pooled analysis of six prospective cohorts using compositional analysis. Br J Sports Med. 2021 Nov;55(22):1277-1285. doi: 10.1136/bjsports-2020-102345. Epub 2021 May 18. PMID 34006506
- [Background] Rodriguez-Gomez I, Manas A, Losa-Reyna J, Rodriguez-Manas L, Chastin SFM, Alegre LM, Garcia-Garcia FJ, Ara I. Associations between sedentary time, physical activity and bone health among older people using compositional data analysis. PLoS One. 2018 Oct 22;13(10):e0206013. doi: 10.1371/journal.pone.0206013. eCollection 2018. PMID 30346973
- [Background] Berkemeyer K, Wijndaele K, White T, Cooper AJ, Luben R, Westgate K, Griffin SJ, Khaw KT, Wareham NJ, Brage S. The descriptive epidemiology of accelerometer-measured physical activity in older adults. Int J Behav Nutr Phys Act. 2016 Jan 7;13:2. doi: 10.1186/s12966-015-0316-z. PMID 26739758
- [Background] Micklesfield LK, Westgate K, Smith A, Kufe CN, Mendham AE, Lindsay T, Wijndaele K, Goedecke JH, Brage S. Physical Activity Behaviors of a Middle-Age South African Cohort as Determined by Integrated Hip and Thigh Accelerometry. Med Sci Sports Exerc. 2022 Sep 1;54(9):1493-1505. doi: 10.1249/MSS.0000000000002940. Epub 2022 Apr 22. PMID 35658390
- [Background] White T, Westgate K, Wareham NJ, Brage S. Estimation of Physical Activity Energy Expenditure during Free-Living from Wrist Accelerometry in UK Adults. PLoS One. 2016 Dec 9;11(12):e0167472. doi: 10.1371/journal.pone.0167472. eCollection 2016. PMID 27936024
- [Background] Dugas LR, Harders R, Merrill S, Ebersole K, Shoham DA, Rush EC, Assah FK, Forrester T, Durazo-Arvizu RA, Luke A. Energy expenditure in adults living in developing compared with industrialized countries: a meta-analysis of doubly labeled water studies. Am J Clin Nutr. 2011 Feb;93(2):427-41. doi: 10.3945/ajcn.110.007278. Epub 2010 Dec 15. PMID 21159791
- [Background] Dowd KP, Szeklicki R, Minetto MA, Murphy MH, Polito A, Ghigo E, van der Ploeg H, Ekelund U, Maciaszek J, Stemplewski R, Tomczak M, Donnelly AE. A systematic literature review of reviews on techniques for physical activity measurement in adults: a DEDIPAC study. Int J Behav Nutr Phys Act. 2018 Feb 8;15(1):15. doi: 10.1186/s12966-017-0636-2. PMID 29422051
- [Background] Schoeller DA. Measurement of energy expenditure in free-living humans by using doubly labeled water. J Nutr. 1988 Nov;118(11):1278-89. doi: 10.1093/jn/118.11.1278. PMID 3142975
- [Background] Prince SA, Adamo KB, Hamel ME, Hardt J, Connor Gorber S, Tremblay M. A comparison of direct versus self-report measures for assessing physical activity in adults: a systematic review. Int J Behav Nutr Phys Act. 2008 Nov 6;5:56. doi: 10.1186/1479-5868-5-56. PMID 18990237
- [Background] Helmerhorst HJ, Brage S, Warren J, Besson H, Ekelund U. A systematic review of reliability and objective criterion-related validity of physical activity questionnaires. Int J Behav Nutr Phys Act. 2012 Aug 31;9:103. doi: 10.1186/1479-5868-9-103. PMID 22938557
- [Background] Hulen E, Ervin A, Schue A, Evans-Young G, Saha S, Yelin EH, Barton JL. Patient goals in rheumatoid arthritis care: A systematic review and qualitative synthesis. Musculoskeletal Care. 2017 Dec;15(4):295-303. doi: 10.1002/msc.1173. Epub 2016 Dec 14. PMID 27976535
- [Background] Axford J, Heron C, Ross F, Victor CR. Management of knee osteoarthritis in primary care: pain and depression are the major obstacles. J Psychosom Res. 2008 May;64(5):461-7. doi: 10.1016/j.jpsychores.2007.11.009. PMID 18440398
- [Background] Cabanas-Sanchez V, Esteban-Cornejo I, Garcia-Esquinas E, Ortola R, Ara I, Rodriguez-Gomez I, Chastin SFM, Rodriguez-Artalejo F, Martinez-Gomez D. Cross-sectional and prospective associations of sleep, sedentary and active behaviors with mental health in older people: a compositional data analysis from the Seniors-ENRICA-2 study. Int J Behav Nutr Phys Act. 2021 Sep 16;18(1):124. doi: 10.1186/s12966-021-01194-9. PMID 34530862
- [Background] Dempsey PC, Aadland E, Strain T, Kvalheim OM, Westgate K, Lindsay T, Khaw KT, Wareham NJ, Brage S, Wijndaele K. Physical activity intensity profiles associated with cardiometabolic risk in middle-aged to older men and women. Prev Med. 2022 Mar;156:106977. doi: 10.1016/j.ypmed.2022.106977. Epub 2022 Feb 4. PMID 35131206
- [Background] Ekelund U, Tarp J, Fagerland MW, Johannessen JS, Hansen BH, Jefferis BJ, Whincup PH, Diaz KM, Hooker S, Howard VJ, Chernofsky A, Larson MG, Spartano N, Vasan RS, Dohrn IM, Hagstromer M, Edwardson C, Yates T, Shiroma EJ, Dempsey P, Wijndaele K, Anderssen SA, Lee IM. Joint associations of accelero-meter measured physical activity and sedentary time with all-cause mortality: a harmonised meta-analysis in more than 44 000 middle-aged and older individuals. Br J Sports Med. 2020 Dec;54(24):1499-1506. doi: 10.1136/bjsports-2020-103270. PMID 33239356
- [Background] Chastin SF, Palarea-Albaladejo J, Dontje ML, Skelton DA. Combined Effects of Time Spent in Physical Activity, Sedentary Behaviors and Sleep on Obesity and Cardio-Metabolic Health Markers: A Novel Compositional Data Analysis Approach. PLoS One. 2015 Oct 13;10(10):e0139984. doi: 10.1371/journal.pone.0139984. eCollection 2015. PMID 26461112
- [Background] Garcia L, Pearce M, Abbas A, Mok A, Strain T, Ali S, Crippa A, Dempsey PC, Golubic R, Kelly P, Laird Y, McNamara E, Moore S, de Sa TH, Smith AD, Wijndaele K, Woodcock J, Brage S. Non-occupational physical activity and risk of cardiovascular disease, cancer and mortality outcomes: a dose-response meta-analysis of large prospective studies. Br J Sports Med. 2023 Aug;57(15):979-989. doi: 10.1136/bjsports-2022-105669. Epub 2023 Feb 28. PMID 36854652
- [Background] Lindsay T, Wijndaele K, Westgate K, Dempsey P, Strain T, De Lucia Rolfe E, Forouhi NG, Griffin S, Wareham NJ, Brage S. Joint associations between objectively measured physical activity volume and intensity with body fatness: the Fenland study. Int J Obes (Lond). 2022 Jan;46(1):169-177. doi: 10.1038/s41366-021-00970-8. Epub 2021 Sep 30. PMID 34593963
- [Background] Strain T, Wijndaele K, Dempsey PC, Sharp SJ, Pearce M, Jeon J, Lindsay T, Wareham N, Brage S. Wearable-device-measured physical activity and future health risk. Nat Med. 2020 Sep;26(9):1385-1391. doi: 10.1038/s41591-020-1012-3. Epub 2020 Aug 17. PMID 32807930
- [Background] Toots A, Rosendahl E, Lundin-Olsson L, Nordstrom P, Gustafson Y, Littbrand H. Usual gait speed independently predicts mortality in very old people: a population-based study. J Am Med Dir Assoc. 2013 Jul;14(7):529.e1-6. doi: 10.1016/j.jamda.2013.04.006. Epub 2013 May 23. PMID 23706405
- [Background] Cleveland RJ, Callahan LF. Can Osteoarthritis Predict Mortality? N C Med J. 2017 Sep-Oct;78(5):322-325. doi: 10.18043/ncm.78.5.322. PMID 28963268
- [Background] Strand V, Wright GC, Bergman MJ, Tambiah J, Taylor PC. Patient Expectations and Perceptions of Goal-setting Strategies for Disease Management in Rheumatoid Arthritis. J Rheumatol. 2015 Nov;42(11):2046-54. doi: 10.3899/jrheum.140976. Epub 2015 Aug 1. PMID 26233504

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT06883591/Prot_SAP_ICF_000.pdf